CLINICAL TRIAL: NCT05352399
Title: Artificial Intelligence + Care Coach Intervention for Persons Living With Dementia and Caregivers
Brief Title: Artificial Intelligence + Care Coach Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Emergency Medicine Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000032226
Record Dates: First submitted 2022-04-18; First posted 2022-04-28 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Dementia; Caregiver; Emergency Department; Artificial Intelligence; Care Transition
MeSH Terms: conditions — Dementia; Emergencies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (NeuViCare AI) (Experimental): An anticipated 55 participants will be part of the Intervention arm participants and will engage with NeuViCare AI, including all variations of its 5 components described further below.
  Interventions: Other: NeuViCare application

INTERVENTIONS:
Other: NeuViCare application — Intervention arm participants will engage with NeuViCare AI, including all variations of its 5 components: 1) NeuViCare Planner - enables review of ordered tests and external resources recommended by the care provider; 2) NeuViCare Task-Support Service - provides context-sensitive, personalized text-based assistance to help patients' complete care plan captured in the NeuViCare Planner; 3) NeuViCare Resource Advisor - presents trusted, unbiased advice to locate nearby resources listed within their care plan; 4) NeuViCare Advisor - educates and trains Persons Living With Dementia (PLWD) and their care partners at the moment of need; and 5) NeuViCare Community Hub - a safe virtual space which enables care partners to interact with other peer care partners to gain their experiential knowledge and emotional support.

SUMMARY:
The purpose of this research study is to develop and test an artificial intelligence intervention for emergency department (ED) discharge care transitions experienced by caregivers of older adults with cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* age ≥65 years with a diagnosis of dementia within the electronic health record OR new cognitive impairment identified during an ED visit
* be fluent in English or Spanish
* discharge after an ED visit
* possession of a smart device (either a phone, tablet, or computer) that has internet access to utilize and interact with NeuViCare AI services

Exclusion Criteria:

- evidence of delirium, by the 4-AT screening tool

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Gettel, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a caregiver-focused study. Although both persons living with cognitive impairment (PLWCI) and their care partners were approached during the recruitment process, only care partners were considered enrolled participants. All baseline and outcome measures, including self-efficacy and burden assessments, were collected solely from enrolled care partners.
  The reported enrollment number and participant flow reflect the number of care partners enrolled, not the number of dyads or PLWCI. No s
Groups:
- Intervention (NeuViCare AI): Participants will be part of the Intervention arm participants and will engage with NeuViCare AI, including all variations of its 5 components described further below.
  NeuViCare application: Intervention arm participants will engage with NeuViCare AI, including all variations of its 5 components: 1) NeuViCare Planner - enables review of ordered tests and external resources recommended by the care provider; 2) NeuViCare Task-Support Service - provides context-sensitive, personalized text-based assistance to help patients' complete care plan captured in the NeuViCare Planner; 3) NeuViCare Resource Advisor - presents trusted, unbiased advice to locate nearby resources listed within their care plan; 4) NeuViCare Advisor - educates and trains Persons Living With Dementia (PLWD) and their care partners at the moment of need; and 5) NeuViCare Community Hub - a safe virtual space which enables care partners to interact with other peer care partners to gain their experiential knowledge and emotional support.
Period: Overall Study
Arm/Group | Intervention (NeuViCare AI)
Started | 40
Completed (34 completed the intervention) | 34
Not Completed | 6
Not completed — Discontinued intervention | 6

BASELINE CHARACTERISTICS:
Arm/Group | Intervention (NeuViCare AI)
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.3 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 26
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 40
Marital Status [Count of Participants; unit: Participants]
  Married | 20
  Divorced | 4
  Single | 4
  Widowed | 12
Form of cognitive impairment [Count of Participants; unit: Participants]
  Diagnosed dementia | 24
  Absence of dementia based on dementia screening score ≥ 2 | 16
Median number of chronic conditions [Median (Inter-Quartile Range); unit: conditions] | 3 [2 to 4]
Emergency Department chief complaint (Most common three) [Count of Participants; unit: Participants]
  Fall | 7
  Altered mental state | 6
  Syncope | 5
Living Situation [Count of Participants; unit: Participants]
  Own home | 10
  With care partner | 30

OUTCOME MEASURES:

1. Primary Outcome: Intervention Appropriateness Measure
Description: Appropriateness is defined as the perceived fit, relevance, or compatibility of the innovation for a given setting or consumer, and/or perceived fit of the innovation to address a particular issue or problem. The measure consists of 4 questions, with an overall score range of 4-20 (higher scores suggest increased appropriateness). Administration time is 1-2 minutes. Measured by survey.
Time Frame: Day 7 and 30
Population: Data presented here is for all caregiver participants that completed the surveys at each time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (NeuViCare AI)
Number analyzed (Participants) | 26
score on a scale
  Day 7: number analyzed (Participants) | 25
  Day 7 | 15.1 (3.6)
  Day 30 | 15.8 (3.9)

2. Primary Outcome: Feasibility of Intervention Measure
Description: Feasibility is defined as the extent to which a new innovation can be successfully used or carried out within a given setting. The measure consists of 4 questions, with an overall score range of 4-20 (higher scores suggest increased feasibility). Administration time is 1-2 minutes. Measured by survey.
Time Frame: Day 7 and 30
Population: Data presented here is for all caregiver participants that completed the surveys at each time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (NeuViCare AI)
Number analyzed (Participants) | 26
score on a scale
  Day 7: number analyzed (Participants) | 25
  Day 7 | 15.1 (3.1)
  Day 30 | 15.5 (3.6)

3. Primary Outcome: Acceptability of Intervention Measure
Description: Acceptability is defined as the perception that a given innovation is agreeable, palatable, or satisfactory. The measure consists of 4 questions, with an overall score range of 4-20 (higher scores suggest increased acceptability). Administration time is 1-2 minutes. Measured by survey.
Time Frame: Day 7 and 30
Population: Data presented here is for all caregiver participants that completed the surveys at each time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (NeuViCare AI)
Number analyzed (Participants) | 26
score on a scale
  Day 7: number analyzed (Participants) | 25
  Day 7 | 15.9 (3.2)
  Day 30 | 15.8 (3.9)

4. Primary Outcome: System Usability Scale
Description: Usability encapsulates several aspects including subjective component assessments of effectiveness, efficiency, and satisfaction. The System Usability Scale consists of 10 questions on effectiveness, efficiency, and satisfaction, with an overall score range of 10-50 (higher scores suggest increased usability). Administration time is 3-5 minutes. Measured by survey.
Time Frame: Day 7 and 30
Population: Data presented here is for all caregiver participants that completed the surveys at each time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (NeuViCare AI)
Number analyzed (Participants) | 26
score on a scale
  Day 7: number analyzed (Participants) | 25
  Day 7 | 30.1 (3.8)
  Day 30 | 29.7 (3.7)

5. Secondary Outcome: Quality of Life (QOL) in Alzheimer's Disease (AD) Scale (QOL-AD)
Description: Total score range 13-52; higher scores indicate better QOL.
Time Frame: Day 0, 7 and 30
Population: Data presented here is for all caregiver participants that completed the surveys at each time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (NeuViCare AI)
Number analyzed (Participants) | 40
score on a scale
  Day 0 | 40.5 (7.4)
  Day 7: number analyzed (Participants) | 25
  Day 7 | 33.8 (9.2)
  Day 30: number analyzed (Participants) | 26
  Day 30 | 36.6 (8)

6. Secondary Outcome: Dyadic Relationship Scale (DRS)
Description: DRS to measure strain between the caregiver and recipient within the last 30 days. Total score range 4-20. High scores indicate high levels of strain.
Time Frame: Day 0, 7 and 30
Population: Data presented here is for all caregiver participants that completed the surveys at each time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (NeuViCare AI)
Number analyzed (Participants) | 40
score on a scale
  Day 0 | 10.7 (3.9)
  Day 7: number analyzed (Participants) | 25
  Day 7 | 10.4 (2.6)
  Day 30: number analyzed (Participants) | 26
  Day 30 | 10.8 (3.5)

7. Secondary Outcome: Zarit Caregiver Burden Scale
Description: The Zarit Caregiver Burden Scale consists of 4 items with the total score ranging between 0-16. Higher scores indicate greater burden. Administration time is approximately 10-15 minutes. Measured by survey.
Time Frame: Day 0, 7 and 30
Population: Data presented here is for all caregiver participants that completed the surveys at each time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (NeuViCare AI)
Number analyzed (Participants) | 40
score on a scale
  Day 0 | 9.2 (4.3)
  Day 7: number analyzed (Participants) | 25
  Day 7 | 9 (2.1)
  Day 30: number analyzed (Participants) | 26
  Day 30 | 8.2 (3.7)

8. Secondary Outcome: Fortinsky Caregiver Self-Efficacy Scale
Description: Used to evaluate the coping ability of daily living. The measure has a total score range from 10-100, with higher scores representing greater self-efficacy. Administration time is approximately 3-5 minutes. Measured by survey.
Time Frame: Day 0, 7, and 30
Population: Data presented here is for all caregiver participants that completed the surveys at each time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (NeuViCare AI)
Number analyzed (Participants) | 40
score on a scale
  Day 0 | 52 (26.3)
  Day 7: number analyzed (Participants) | 25
  Day 7 | 57.6 (23.1)
  Day 30: number analyzed (Participants) | 26
  Day 30 | 65.8 (17.8)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Intervention (NeuViCare AI)
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT05352399/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT05352399/ICF_001.pdf